CLINICAL TRIAL: NCT06245980
Title: Role of SGLT2I in Diabetic Patients With Myocardial Infarction
Brief Title: Role of SGLT2I in Patients With Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dongying Zhang (Other)
Responsible Party: Sponsor-Investigator, Dongying Zhang, Professor, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: 20230515
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-05

CONDITIONS: Myocardial Infarction; Diabetes Mellitus
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With SGLT2I
  Interventions: Drug: SGLT2 inhibitor
- Without SGLT2i

INTERVENTIONS:
Drug: SGLT2 inhibitor — According to whether SGLT2i was used
  Groups: With SGLT2I

SUMMARY:
Role of sglt2I in diabetic patients with myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

1. Acute myocardial infarction patients
2. Type 2 diabetics.

Exclusion Criteria:

1. Patients undergoing coronary artery bypass grafting (CABG).
2. Severe valvular heart disease.
3. Contraindications of secondary medical preventive therapy for myocardial infarction, such as β-blockers, angiotensin-converting enzyme inhibitors (ACEI)/ angiotensin-converting enzyme inhibitors (ARBs), antiplatelets, and statins.
4. Previously used SGLT2i.
5. Severe hepatic and renal insufficiency.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myocardial infarction patients with diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 24months
  cardiovascular death and heart failure and myocardial infarction
Heart failure readmission | 24months
  Heart failure readmission

SECONDARY OUTCOMES:
Recurrent myocardial infarction | 24months
  Recurrent myocardial infarction
cardiovascular death | 24months
  cardiovascular death

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Luo S, Liu H, Li Z, Zhou Y, He S, Zhang D, Qin S, Wen X. Effects of SGLT2 Inhibitor in Patients with Diabetes with Newly Diagnosed Acute Myocardial Infarction: A Multicenter Prospective Cohort Study. Cardiovasc Drugs Ther. 2025 May 22. doi: 10.1007/s10557-025-07716-y. Online ahead of print. PMID 40402390